CLINICAL TRIAL: NCT00202306
Title: An Open-labeled, Parallel-group, Single-blinded (Rater) Pilot Study to Investigate the Neuroprotective Effects of of Low-dose Lithium in Young Subjects at Ultra High Risk (UHR) of Developing a First-episode Psychotic Disorder
Brief Title: Indicated Prevention of Psychotic Disorders With Low-dose Lithium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Gregor Berger MD, Senior Lecturer, ORYGEN Research Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRI 01-038; E/01/028
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Bipolar Disorder; Psychotic Disorders
Keywords: at risk mental state; prodrome; ultra high risk; first episode psychosis; schizophrenia; bipolar disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lithium carbonate

SUMMARY:
This study investigates the neuroprotective properties of low-dose lithium in young individuals at ultra-high risk of developping a first psychotic episode. Fourty individuals having some symptoms of an emerging psychotic disorders (without meeting the threshold for a full-blown mental illness) will be treated with a low dose of lithium (about a third of the dose that is usually used to treat acute mania). We will assess the progression of the conditions of these individuals on a montly bases for a year. We will do behavioural, cognitive and imaging assessments prior start of the treatment, after three months and one year. We hope to demonstrate that low dose lithium will stop or even reverse the progression of disease. We expect that behavioral, cognitive and in vivo brain imaging parameters in those individuals treated with low dose lithium improve, compared to the monitoring group.

DETAILED DESCRIPTION:
To investigate whether low-dose lithium is an effective agent in indicated prevention amongst subjects at ultra-high risk of developing a psychotic disorder. This aim will be achieved by treating a high-risk patient population with low-dose lithium (450mg/day) and investigating its effects using clinical, neuropsychological, neuroimaging and cell biological approaches. We will recruit 30 patients considered to be at ultra-high risk of developing a first psychotic episode, currently receiving treatment at the Personal Assessment and Crisis Evaluation (PACE) clinic in Melbourne, Australia. PACE criteria for identifying patients at high risk include subjects with a family history of psychosis and a decrease in functioning (30% GAF) AND/OR attenuated psychotic symptoms AND/OR brief psychotic symptoms (BLIPS) resolving without treatment. Patients who give informed consent will receive treatment with a slow release form of low dose lithium for a period of a year, plus supportive therapy. Patients who do not consent will receive supportive therapy only. Assessments will be conducted at baseline, twelve weeks and one year post-recruitment. Assessments will include cognitive functioning, structural MRI, 1H-MRS at 3Tesla and cell biological parameters (bcl-2, AP-1; NIMH, Washington DC). In addition, all patients will be seen on a monthly basis for a clinical interview, covering psychopathology, global functioning, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Attenuated psychotic symptoms
* Self-limited brief psychotic episode
* Family History of psychosis and decrease in functioning over last year

Exclusion Criteria:

* Organic causes of subthreshold psychotic symptoms (eg. epilepsy)
* More than one week of neuroleptic treatment

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement
Cognitive improvement
Brain structural change (grey matter, ventricle to brain ratio)
Brain metabolic changes (Proton Magnetic Resonance Spectroscopy)

SECONDARY OUTCOMES:
Transition rate to Psychosis
Quality of life
serum apoptosis parameters (eg. bcl2)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor E Berger, MD, Principal Investigator — University of Melbourne, Department of Psychiatry, ORYGEN Research Centre
Locations (1):
- ORYGEN Youth Health, PACE Clinic, Parkville, Victoria, Australia

REFERENCES:
- [Background] Berger GE, Wood S, McGorry PD. Incipient neurovulnerability and neuroprotection in early psychosis. Psychopharmacol Bull. 2003 Spring;37(2):79-101. PMID 14566217
- See also: Description of Unit of Neuroprotection in Young People (UNYP) — http://www.ORYGEN.org.au